CLINICAL TRIAL: NCT01685008
Title: A Phase IIa, Open-label, Multicenter Study of Single-agent MOR00208, an Fc-optimized Anti-CD19 Antibody, in Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: Study of Fc-Optimized Anti-CD19 Antibody (MOR00208) to Treat Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR208C201; 2012-002659-41 (EudraCT Number)
Record Dates: First submitted 2012-09-03; First posted 2012-09-13 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: NHL; CD19; MOR208; MOR00208; Xmab5574; B-Cell Non-Hodgkin´s Lymphoma; Fc-optimized Anti-CD19 Antibody; Tafasitamab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tafasitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MOR00208 (formerly Xmab5574) (Experimental): intravenous Infusion of MOR00208, Fc-Optimized Anti-CD19 Antibody
  Interventions: Drug: MOR00208 (formerly Xmab 5574)

INTERVENTIONS:
Drug: MOR00208 (formerly Xmab 5574)
  Other Names: MOR208

SUMMARY:
This is an open-label, multicenter study to characterize the safety and efficacy of the human anti-CD19 antibody MOR00208 in adult patients with relapsed/refractory non-Hodgkin's lymphoma (NHL) who have received at least 1 prior therapy containing rituximab (at least once).

DETAILED DESCRIPTION:
The study enrols patients from four different NHL subtypes: follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma (MCL) and other indolent NHL (iNHL). The study will employ a two-stage design where the decision to further enrol any NHL subtype in stage 2 will depend on best responses after two or three cycles in stage 1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Histologically-confirmed diagnosis according to Revised European American Lymphoma/World Health Organization classification, of the following B-cell lymphomas:

   1. FL
   2. Other indolent NHL (eg, MZL/MALT)
   3. DLBCL
   4. MCL
3. Patients' NHL must have progressed after at least 1 prior rituximab containing regimen.
4. One site of measurable disease by magnetic resonance imaging (MRI) or computed tomography (CT) scan defined as at least one lesion that measures at least 1.5 × 1.5 cm.

   Exception:

   For patients with MCL only, patients with nonmeasurable disease but evaluable sites (bone marrow, spleen, peripheral blood, gastrointestinal tract) can be enrolled.
5. Patients who have previously received an autologous stem cell transplantation must be at least 4 weeks post-transplant before study drug administration and must have exhibited a full haematological recovery.
6. Discontinued previous monoclonal antibody therapy (except rituximab) or radioimmunotherapy administration for at least 60 days before study drug administration.
7. Off rituximab for at least 14 days before the screening visit and be confirmed to have either no response or have disease progression after rituximab treatment.
8. Patients with DLBCL had a positive [18F]fluorodeoxyglucose-positron emission tomography (FDG-PET) scan at baseline (Cheson 2007 response criteria).
9. Life expectancy of > 3 months.
10. Eastern Cooperative Oncology Group (ECOG) performance status of < 3.
11. Laboratory criteria at screening:

    1. Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L
    2. Platelet count ≥ 75 × 10^9/L without previous transfusion within 10 days of first study drug administration
    3. Haemoglobin ≥ 8.0 g/dL (may have been transfused)
    4. Serum creatinine < 2.0 x upper limit of normal (ULN)
    5. Total bilirubin ≤ 2.0 × ULN
    6. Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN
12. If a female of childbearing potential, a negative pregnancy test must be confirmed before enrolment and use of double-barrier contraception or oral contraceptive plus barrier contraceptive must be used during the study and for 3 months after the last dose, or confirmation of having undergone clinically documented total hysterectomy and/or oophorectomy, tubal ligation.
13. If a male, an effective barrier method of contraception must be used during the study and for 3 months after the last dose if the patient is sexually active with a female of childbearing potential.
14. Able to comply with all study-related procedures, medication use, and evaluations.
15. Able to understand and give written informed consent and comply with the study protocol.

Exclusion Criteria:

1. Previous treatment with cytotoxic chemotherapy, immunotherapy, radiotherapy or other lymphoma specific therapy within 14 days before the screening visit or patient has not recovered from side effects of previous lymphoma-specific therapy.
2. Treatment with a systemic investigational agent within 28 days before the screening visit.
3. Previous treatment with an anti-CD19 antibody or fragments.
4. Previous allogenic stem cell transplantation.
5. Known or suspected hypersensitivity to the excipients contained in the study drug formulation.
6. Clinically significant cardiovascular disease or cardiac insufficiency, cardiomyopathy, preexisting clinically significant arrhythmia, acute myocardial infarction within 3 months of enrolment, angina pectoris within 3 months of enrolment.
7. Patients with positive hepatitis serology:

   Hepatitis B (HBV): Patients with positive serology for HBV defined as positivity for hepatitis B surface antigen (HBsAg) or total anti-hepatitis B core antibody (anti-HBc). Patients positive for anti-HBc may be included if HBV DNA is not detectable.

   Hepatitis C (HCV): Patients positive HCV serology (defined as positive for anti-HCV antibody [anti-HCV]) unless HCV-ribonucleic acid (RNA) is confirmed negative.
8. History of HIV infection.
9. Any active systemic infection (viral, fungal, or bacterial) requiring active parenteral antibiotic therapy within 4 weeks of study drug administration.
10. Current treatment with immunosuppressive agents other than prescribed corticosteroids (not more than 10-mg prednisone equivalent).
11. Major surgery or radiation therapy within 4 weeks before first study drug administration.
12. Systemic diseases (cardiovascular, renal, hepatic, etc) that would prevent study treatment in the investigator's opinion.
13. History or clinical evidence of central nervous system (CNS), meningeal, or epidural disease, including brain metastasis.
14. Active treatment/chemotherapy for another primary malignancy within the past 5 years (except for ductal breast cancer in situ, non-melanoma skin cancer, prostate cancer not requiring treatment, and cervical carcinoma in situ).
15. Pregnancy or breastfeeding in women and women of childbearing potential not using an acceptable method of birth control.
16. History of noncompliance to medical regimens or patients who are considered potentially unreliable not cooperative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (4):
  - MorphoSys Research Site, Norwalk, Connecticut
  - MorphoSys Research Site, Hackensack, New Jersey
  - Morphosys Research Site, Columbus, Ohio
  - Morphosys Research Site, Lubbock, Texas
- Belgium (2):
  - MorphoSys Research Site, Brussels
  - MorphoSys Research Site, Edegem
- Germany (3):
  - MorphoSys Research Site, Berlin
  - MorphoSys Research Site, Mainz
  - Morphosys Research Site, Ulm
- Hungary (2):
  - Morphosys Research Site, Budapest
  - Morphosys Research Site, Debrecen
- Italy (5):
  - MorphoSys Research Site, Bologna
  - MorphoSys Research Site, Florence
  - Morphosys, Genova
  - Morphosys Research Site, Modena
  - Morphosys Research Site, Novara
- Poland (4):
  - MorphoSys Research Site, Chorzów
  - Morphosys Research Site, Krakow
  - Morphosys Research Site, Lódz
  - MorphoSys Research Site, Słupsk
- Spain (2):
  - Morphosys Research Site, Madrid
  - Morphosys Research Site, Seville

REFERENCES:
- [Derived] Jurczak W, Zinzani PL, Gaidano G, Goy A, Provencio M, Nagy Z, Robak T, Maddocks K, Buske C, Ambarkhane S, Winderlich M, Dirnberger-Hertweck M, Korolkiewicz R, Blum KA. Phase IIa study of the CD19 antibody MOR208 in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma. Ann Oncol. 2018 May 1;29(5):1266-1272. doi: 10.1093/annonc/mdy056. PMID 29444231

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients who fulfilled all the inclusion criteria and none of the exclusion criteria were enrolled and received MOR00208 infusion. Per planned analyses, patient disposition and treatment discontinuation is summarized by NHL subtype.
Groups:
- FL Subtype: Patients with follicular lymphoma. All patients received 12 mg/kg MOR00208 administered as an intravenous infusion.
- DLBCL Subtype: Patients with diffuse large B-cell lymphoma. All patients received 12 mg/kg MOR00208 administered as an intravenous infusion.
- MCL Subtype: Patients with mantle cell lymphoma. All patients received 12 mg/kg MOR00208 administered as an intravenous infusion.
- Other iNHL: Patients with other indolent non-Hodgkin's lymphoma. All patients received 12 mg/kg MOR00208 administered as an intravenous infusion.
Period: Main Study Treatment (Cycles 1 - 2)
Arm/Group | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL
Started | 34 | 35 | 12 | 11
Completed (Patients were considered to have completed the study if they finished the first 2 cycles of treatment plus the end of cycle 2 assessments.) | 30 | 25 | 10 | 10
Not Completed | 4 | 10 | 2 | 1
Not completed — Adverse Event | 2 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 2 | 4 | 1 | 0
Not completed — Death | 0 | 3 | 1 | 0
Period: Cycle 3 and Maintenance Treatment
Arm/Group | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL
Started (Includes all patients that completed the first 2 cycles of treatment.) | 30 | 25 | 10 | 10
Began Cycle 3 Treatment | 25 | 13 | 5 | 7
Entered Maintenance Phase Treatment | 8 | 6 | 0 | 2
Completed | 0 | 1 | 0 | 0
Not Completed | 30 | 24 | 10 | 10

BASELINE CHARACTERISTICS:
Population: Per planned analyses, baseline characteristics are summarized by NHL subtype.
Groups:
- Total: Total of all reporting groups
Arm/Group | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | Total
Number analyzed (Participants) | 34 | 35 | 12 | 11 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 6 | 2 | 43
  >=65 years | 15 | 19 | 6 | 9 | 49
Age, Continuous [Mean (Full Range); unit: years] | 62.88 [40 to 87] | 66.71 [35 to 90] | 64.92 [56 to 74] | 70.91 [45 to 83] | 65.57 [35 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 1 | 6 | 36
  Male | 16 | 24 | 11 | 5 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 32 | 33 | 11 | 11 | 87
  Other | 2 | 1 | 0 | 0 | 3
Height [Mean (Full Range); unit: cm] — Population: Height was not collected at Screening for 2 patients (minor protocol noncompliance)
  cm
    number analyzed (Participants) | 34 | 33 | 12 | 11 | 90
    (all) | 170.26 [150 to 244] | 168.24 [150 to 184] | 171.00 [150 to 191] | 167.64 [160 to 178] | 169.30 [150 to 244]
Weight [Mean (Full Range); unit: kg] | 78.62 [51.0 to 123.6] | 75.52 [46.0 to 122.5] | 82.52 [63.9 to 131.0] | 71.53 [50.0 to 92.0] | 77.10 [46.0 to 131.0]
BMI [Mean (Full Range); unit: kg/m^2] — Population: Height was not collected at Screening for 2 patients (minor protocol noncompliance)
  kg/m^2
    number analyzed (Participants) | 34 | 33 | 12 | 11 | 90
    (all) | 27.26 [12.6 to 39.3] | 26.52 [18.9 to 41.1] | 28.03 [22.1 to 36.1] | 25.36 [18.4 to 32.0] | 26.86 [12.6 to 41.1]
NHL Subtype [Count of Participants; unit: Participants]
  Follicular lymphoma | 34 | 0 | 0 | 0 | 34
  Diffuse large B-cell lymphoma | 0 | 35 | 0 | 0 | 35
  Mantle cell lymphoma | 0 | 0 | 12 | 0 | 12
  Other indolent NHL | 0 | 0 | 0 | 11 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Proportion of patients with Complete Remission (CR; disappearance of all evidence of disease) or Partial Remission (PR; regression of measurable disease and no new sites), assessed as per the 2007 International Working Group (IWG) response criteria by radiographic evaluations (CT, PET, MRI, or other).
Time Frame: From first dose until Follow-up Visit 12, up to 4.5 years
Population: The Intent-to-treat (ITT) Population consisted of all patients who received at least one dose of study drug. Patients without any post-Baseline assessment of NHL response were included as non-responders. Per pre-specified analysis plan, efficacy analyses are summarized overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Count of Participants; unit: Participants
Groups:
- Total: All patients received 12 mg/kg MOR00208 administered as an intravenous infusion.
- FL + Other iNHL: Combined group of patients with follicular lymphoma and patients with other indolent non-Hodgkin's lymphoma. All patients received 12 mg/kg MOR00208 administered as an intravenous infusion.
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 92 | 34 | 35 | 12 | 11 | 45
Participants
  Complete remission | 6 | 2 | 2 | 0 | 2 | 4
  Partial remission | 16 | 8 | 7 | 0 | 1 | 9

2. Secondary Outcome: Stable Disease (SD) Rate
Description: Proportion of patients with Stable Disease (failure to attain CR/PR with no progressive disease)
Time Frame: From first dose until Follow-up Visit 12, up to 4.5 years
Population: The ITT Population consisted of all patients who received at least one dose of study drug. Patients without any post-Baseline assessment of NHL response were included as non-responders. Per pre-specified analysis plan, efficacy analyses are summarized overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 92 | 34 | 35 | 12 | 11 | 45
Participants | 31 | 16 | 5 | 6 | 4 | 20

3. Secondary Outcome: Duration of Response (DoR)
Description: Time from first CR or PR to first documentation of relapse/progression (any new lesion or increase by ≥ 50% of previously identified site)
Time Frame: From first dose until Follow-up Visit 12, up to 4.5 years
Population: Patients in the ITT Population who had any response (CR or PR) during the study. Per pre-specified analysis plan, efficacy analyses are summarized overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 22 | 10 | 9 | 0 | 3 | 13
months | 24.0 [11.1 to NA] — Patients who showed a response during the study but did not have documented progression (as described in the pre-specified analysis plan) were considered censored. Due to this statistical data censoring, there was an insufficient number of patients with events in the analysis population to compute median and/or confidence interval(s). | 24.0 [2.6 to NA] — Patients who showed a response during the study but did not have documented progression (as described in the pre-specified analysis plan) were considered censored. Due to this statistical data censoring, there was an insufficient number of patients with events in the analysis population to compute median and/or confidence interval(s). | 20.1 [1.1 to NA] — Patients who showed a response during the study but did not have documented progression (as described in the pre-specified analysis plan) were considered censored. Due to this statistical data censoring, there was an insufficient number of patients with events in the analysis population to compute median and/or confidence interval(s). |  | NA [NA to NA] — No responders had documented progression, therefore all patients in this population were censored and no median or confidence intervals were applicable. | NA [3.6 to NA] — Patients who showed a response during the study but did not have documented progression (as described in the pre-specified analysis plan) were considered censored. Due to this statistical data censoring, there was an insufficient number of patients with events in the analysis population to compute median and/or confidence interval(s).

4. Secondary Outcome: Time to Progression (TTP)
Description: Time from first dosing until documentation of progression or death due to lymphoma
Time Frame: From first dose until Follow-up Visit 12, up to 4.5 years
Population: Patients in the ITT Population with documented progression of disease. Per pre-specified analysis plan, efficacy analyses are summarized overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 76 | 31 | 25 | 11 | 9 | 40
months | 5.4 [3.4 to 12.0] | 8.8 [5.4 to 20.5] | 3.1 [2.1 to 15.4] | 3.0 [1.8 to NA] — Patients who did not have documented radiological progression (as described in the pre-specified analysis plan) were considered censored. Due to this statistical data censoring, there was an insufficient number of patients with events in the analysis population to compute median and/or confidence interval(s). | NA [2.0 to NA] — Patients who did not have documented radiological progression (as described in the pre-specified analysis plan) were considered censored. Due to this statistical data censoring, there was an insufficient number of patients with events in the analysis population to compute median and/or confidence interval(s). | 6.6 [5.3 to 20.5]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from first dosing until progression or death due to any case
Time Frame: From first dose until Follow-up Visit 12, up to 4.5 years
Population: Patients in the ITT Population with documented progression of disease or death from any cause. Per pre-specified analysis plan, efficacy analyses are summarized overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 80 | 31 | 28 | 12 | 9 | 40
months | 5.4 [3.2 to 9.9] | 8.8 [5.4 to 20.5] | 2.7 [2.1 to 13.2] | 2.1 [1.7 to NA] — Patients who did not have documented radiological progression, or death occurred beyond a pre-specified time frame (as described in the pre-specified analysis plan) were considered censored. Due to this statistical data censoring, there was an insufficient number of patients with events in the analysis population to compute median and/or confidence interval(s). | NA [2.0 to NA] — Patients who did not have documented radiological progression, or death occurred beyond a pre-specified time frame (as described in the pre-specified analysis plan) were considered censored. Due to this statistical data censoring, there was an insufficient number of patients with events in the analysis population to compute median and/or confidence interval(s). | 6.6 [5.3 to 20.5]

6. Secondary Outcome: Incidence and Severity of Adverse Events (AEs)
Description: Number of patients with treatment-emergent AEs rated Mild, Moderate, and Severe
Time Frame: From first dose until 30 days after last dose of MOR00208, up to 8.5 years
Population: The Safety Population consisted of all patients who received at least one dose of study drug. Per pre-specified analysis plan, adverse event analyses are summarized overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 92 | 34 | 35 | 12 | 11 | 45
Participants
  Mild | 29 | 10 | 12 | 1 | 6 | 16
  Moderate | 20 | 8 | 8 | 2 | 2 | 10
  Severe | 6 | 2 | 4 | 0 | 0 | 2

7. Secondary Outcome: Number and Proportion of Patients Who Potentially Developed Anti-MOR00208 Antibodies and Semiquantitative Anti-MOR00208 Antibody Assessments
Description: Number of patients with at least one positive (+ve) post-Baseline sample containing positive anti-MOR00208 antibodies; Baseline (pre-dose) sample has to be tested negative (-ve)
Time Frame: From first dose until Follow-up Visit 3, up to 7 months
Population: The Safety Population (all patients who received at least one dose of study drug). Per pre-specified analysis plan, statistical summaries are provided overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 92 | 34 | 35 | 12 | 11 | 45
Participants
  Yes (at least 1 +ve post-Baseline sample, including +ve last sample; Baseline must be -ve) | 0 | 0 | 0 | 0 | 0 | 0
  No (Baseline and all post-Baseline samples are -ve) | 82 | 31 | 31 | 10 | 10 | 41
  Transient (at least 1 +ve post-Baseline sample but -ve last sample; Baseline must be -ve) | 0 | 0 | 0 | 0 | 0 | 0
  Not evaluable (pre-dose Baseline sample tested +ve) | 5 | 3 | 1 | 1 | 0 | 3
  Missing (no post-Baseline measurement available) | 5 | 0 | 3 | 1 | 1 | 1

8. Secondary Outcome: Pharmacokinetic (PK) Parameter: Maximum Serum Concentration Observed (Cmax) of MOR00208
Description: The highest concentration of MOR00208 measured in serum
Time Frame: Estimated from first dose (samples taken on first day of dosing at pre-dose, end of infusion, after 1 hour, 4 hours, 24 hours, and pre-dose on Day 8)
Population: The PK Population included all patients who had at least one quantifiable serum MOR00208 concentration. PK parameters were calculated as data permitted. Per pre-specified analysis plan, statistical summaries are provided overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 85 | 33 | 32 | 11 | 9 | 42
μg/mL | 263.1 (111.35) | 276.6 (73.10) | 253.4 (157.79) | 260.0 (69.85) | 251.5 (70.31) | 271.2 (72.42)

9. Secondary Outcome: PK Parameter: Time to Maximum Serum Concentration Observed (Tmax) of MOR00208
Description: The time to highest concentration of MOR00208 measured in serum
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 85 | 33 | 32 | 11 | 9 | 42
hours | 5.8 (17.46) | 4.7 (5.27) | 8.5 (27.99) | 3.0 (1.03) | 3.4 (1.38) | 4.4 (4.72)

10. Secondary Outcome: PK Parameter: Apparent Trough Serum Concentration Before Dosing (Clast) of MOR00208
Description: The last quantifiable concentration from the first dose of MOR00208
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 85 | 33 | 32 | 11 | 9 | 42
μg/mL | 81.0 (36.66) | 88.6 (39.50) | 69.6 (28.96) | 82.4 (34.54) | 92.2 (47.23) | 89.3 (40.69)

11. Secondary Outcome: PK Parameter: Area Under the Concentration Curve From Dose Time Zero to the Time the Last Quantifiable Concentration is Observed (AUC[0-t]) of MOR00208
Description: Area under the concentration curve. The time curve from time zero (0) to the time that the last concentration above the lower limit of quantification (LLQ) is observed.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 85 | 33 | 32 | 11 | 9 | 42
h*μg/mL | 21942.5 (11847.35) | 25088.6 (16245.82) | 19106.3 (8170.03) | 21617.1 (4577.21) | 20888.5 (7669.67) | 24188.6 (14849.65)

12. Secondary Outcome: PK Parameter: Area Under the Concentration Curve From Dose Time Zero to Infinity (AUC[0-inf]) of MOR00208
Description: Area under the concentration curve. The time curve from time zero (0) to infinity (inf), where infinity is computed from AUC0-t + [Ct/λZ)]. Ct is calculated from the concentration at the last sampling time at which the sample is above LLQ.
Time Frame: Estimated from final dose (samples collected on the last day of Cycle 3 [C3D28; each cycle is 28 days long], and Follow-up Visits 1 [C3D28 + 4 weeks], 2 [C3D28 + 10 weeks], and 3 [C3D28 + 16 weeks])
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 91 | 33 | 35 | 12 | 11 | 44
h*μg/mL | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation.

13. Secondary Outcome: PK Parameter: Apparent Terminal Rate Constant (λz) of MOR00208
Description: Apparent terminal rate constant calculated from the regression analysis (slope) from the log-transformed measured concentrations on the terminal phase of the time-point concentration curve
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 12 | 9 | 0 | 2 | 1 | 10
1/h | 0.00214 (0.000665) | 0.00214 (0.000707) |  | 0.00207 (0.000896) | 0.00234 (NA) — Standard deviation is not applicable for a sample size of 1. | 0.00216 (0.000670)

14. Secondary Outcome: PK Parameter: Apparent Terminal Half-life (t[1/2]) of MOR00208
Description: Apparent terminal half-life calculated from ln(2)/λz
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 12 | 9 | 0 | 2 | 1 | 10
days | 14.75111 (4.680075) | 14.87185 (4.863339) |  | 15.42457 (6.690102) | 12.31761 (NA) — Standard deviation is not applicable for a sample size of 1. | 14.61642 (4.655799)

15. Secondary Outcome: PK Parameter: Total Body Clearance (CL) of MOR00208
Description: Total body clearance calculated for single or multiple doses: dose(s)/AUC(0-inf)
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 91 | 33 | 35 | 12 | 11 | 44
L/h | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation.

16. Secondary Outcome: PK Parameter: Apparent Volume of Distribution (Vz) of MOR00208
Description: Apparent volume of distribution during the terminal phase, calculated from dose/(AUC(0-inf)*λz)
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 91 | 33 | 35 | 12 | 11 | 44
L | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation. | NA (NA) — There were not sufficient data available to allow parameter estimation.

17. Secondary Outcome: Absolute Change From Baseline in Measurements of B-cell Populations
Description: Actual change from baseline will be summarized descriptively by visit for the pharmacodynamic parameter: B-cell populations
Time Frame: Cycle 1 Day 1 (Baseline) to Cycle 1: Days 8, 15, and 22; Cycles 2 and 3: Days 1, 15, and 28 (each cycle is 28 days); End of Study (up to 7.5 years)
Population: Pharmacodynamic samples were collected at timepoints through the study where possible. Per pre-specified analysis plan, statistical summaries are provided overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Median (95% Confidence Interval); unit: 10^6 cells/L
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 70 | 26 | 31 | 8 | 5 | 31
10^6 cells/L
  Cycle 1 Day 8: number analyzed (Participants) | 65 | 24 | 28 | 8 | 5 | 29
  Cycle 1 Day 8 | -13.60 [-50.250 to -1.000] | -68.00 [-141.000 to -1.000] | 0.00 [-13.600 to 10.000] | -61.13 [-214.200 to 7618.000] | -65.00 [-108.000 to 13.000] | -65.00 [-108.000 to -2.000]
  Cycle 1 Day 15: number analyzed (Participants) | 65 | 26 | 27 | 7 | 5 | 31
  Cycle 1 Day 15 | -15.00 [-55.940 to -3.000] | -60.50 [-171.000 to -10.000] | -3.00 [-15.000 to 6.000] | -47.00 [-687.000 to 26570.000] | -47.00 [-110.000 to 0.000] | -57.00 [-110.020 to -10.000]
  Cycle 1 Day 22: number analyzed (Participants) | 61 | 23 | 26 | 7 | 5 | 28
  Cycle 1 Day 22 | -14.00 [-57.000 to -4.500] | -34.00 [-148.000 to -6.000] | -4.25 [-19.000 to 0.000] | -65.01 [-680.000 to 1487.000] | -60.00 [-120.000 to 33.000] | -44.00 [-105.980 to -6.000]
  Cycle 2 Day 1: number analyzed (Participants) | 58 | 24 | 24 | 5 | 5 | 29
  Cycle 2 Day 1 | -14.00 [-51.710 to -3.600] | -45.00 [-141.000 to -2.000] | -4.00 [-17.000 to 1.000] | -51.71 [-697.000 to 2025.000] | -3.00 [-121.000 to 42.000] | -34.00 [-116.390 to -2.000]
  Cycle 2 Day 15: number analyzed (Participants) | 54 | 20 | 22 | 7 | 5 | 25
  Cycle 2 Day 15 | -24.00 [-61.000 to -12.000] | -47.50 [-181.210 to 0.000] | -14.25 [-23.000 to -4.900] | -61.45 [-673.000 to 9637.000] | -56.00 [-120.000 to 20.000] | -56.00 [-120.000 to -5.500]
  Cycle 2 Day 28: number analyzed (Participants) | 48 | 21 | 18 | 5 | 4 | 25
  Cycle 2 Day 28 | -27.68 [-59.000 to -8.000] | -28.00 [-115.120 to -0.800] | -14.50 [-35.000 to -1.970] | -176.85 [-661.000 to -28.000] | -38.00 [-120.000 to -4.000] | -28.00 [-94.000 to -3.880]
  Cycle 3 Day 1: number analyzed (Participants) | 33 | 17 | 9 | 3 | 4 | 21
  Cycle 3 Day 1 | -36.00 [-117.990 to 0.000] | -43.00 [-171.000 to 5.000] | -16.00 [-238.000 to 0.000] | -13.06 [-718.000 to 2.000] | -68.00 [-129.000 to 16.000] | -64.00 [-129.000 to 5.000]
  Cycle 3 Day 15: number analyzed (Participants) | 30 | 16 | 8 | 3 | 3 | 19
  Cycle 3 Day 15 | -36.50 [-135.720 to 0.000] | -33.50 [-171.000 to 10.000] | -22.00 [-241.000 to 21.000] | -256.72 [-615.000 to -30.000] | -77.00 [-127.000 to -6.000] | -35.00 [-127.000 to 9.000]
  Cycle 3 Day 28: number analyzed (Participants) | 33 | 18 | 8 | 3 | 4 | 22
  Cycle 3 Day 28 | -46.00 [-94.000 to -8.370] | -60.50 [-171.000 to 10.000] | -16.50 [-124.800 to 35.000] | -43.00 [-689.000 to 76.530] | -59.00 [-129.000 to -5.000] | -60.50 [-121.180 to -5.000]
  Study Completion/Early Termination: number analyzed (Participants) | 43 | 17 | 17 | 5 | 4 | 21
  Study Completion/Early Termination | -15.00 [-69.820 to 4.000] | -72.00 [-241.000 to 8.000] | -1.67 [-22.100 to 7.000] | -49.00 [-618.000 to 63413.000] | -40.50 [-133.000 to 22.000] | -72.00 [-240.000 to 8.000]

18. Secondary Outcome: Percent Change From Baseline in Measurements of B-cell Populations
Description: Relative change from baseline will be summarized descriptively by visit for the pharmacodynamic parameter: B-cell populations
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 70 | 26 | 31 | 8 | 5 | 31
percentage change from baseline
  Cycle 1 Day 8: number analyzed (Participants) | 60 | 22 | 25 | 8 | 5 | 27
  Cycle 1 Day 8 | -42.07 [-70.588 to -2.793] | -80.64 [-95.914 to -25.000] | -0.64 [-49.333 to 72.857] | -40.32 [-77.154 to 1451.048] | -74.47 [-81.203 to 118.182] | -76.47 [-85.116 to -25.000]
  Cycle 1 Day 15: number analyzed (Participants) | 61 | 24 | 25 | 7 | 5 | 29
  Cycle 1 Day 15 | -50.00 [-79.422 to -32.353] | -87.11 [-95.947 to -46.341] | -32.35 [-67.442 to 11.429] | -40.17 [-85.160 to 5060.952] | -50.00 [-87.059 to 0.000] | -82.71 [-94.253 to -46.341]
  Cycle 1 Day 22: number analyzed (Participants) | 57 | 21 | 24 | 7 | 5 | 26
  Cycle 1 Day 22 | -55.88 [-82.625 to -27.500] | -83.23 [-100.000 to -35.800] | -35.77 [-67.857 to -5.714] | -82.62 [-90.556 to 33.514] | -63.83 [-90.226 to 71.739] | -68.39 [-96.279 to -35.800]
  Cycle 2 Day 1: number analyzed (Participants) | 54 | 22 | 22 | 5 | 5 | 27
  Cycle 2 Day 1 | -55.63 [-80.000 to -27.273] | -82.65 [-94.312 to -25.102] | -40.18 [-61.905 to 27.778] | -72.03 [-85.171 to 45.639] | -27.27 [-90.977 to 54.348] | -80.18 [-92.093 to -25.102]
  Cycle 2 Day 15: number analyzed (Participants) | 50 | 18 | 20 | 7 | 5 | 23
  Cycle 2 Day 15 | -73.80 [-83.542 to -57.407] | -81.98 [-100.000 to -35.667] | -67.32 [-83.542 to -31.250] | -74.07 [-93.373 to 217.196] | -71.76 [-100.000 to 43.478] | -78.05 [-97.957 to -57.407]
  Cycle 2 Day 28: number analyzed (Participants) | 45 | 20 | 16 | 5 | 4 | 24
  Cycle 2 Day 28 | -76.47 [-86.458 to -38.095] | -87.25 [-100.000 to -7.143] | -59.07 [-83.415 to -23.529] | -71.67 [-96.062 to -30.769] | -52.89 [-90.226 to -18.085] | -82.87 [-94.419 to -18.085]
  Cycle 3 Day 1: number analyzed (Participants) | 29 | 15 | 7 | 3 | 4 | 19
  Cycle 3 Day 1 | -79.63 [-94.585 to -3.666] | -93.06 [-96.639 to 22.997] | -82.64 [-98.333 to 142.105] | -3.67 [-87.242 to 3.704] | -76.06 [-96.992 to 145.455] | -79.63 [-95.608 to 22.997]
  Cycle 3 Day 15: number analyzed (Participants) | 27 | 14 | 7 | 3 | 3 | 17
  Cycle 3 Day 15 | -72.07 [-93.953 to -33.333] | -76.61 [-96.479 to 48.780] | -45.24 [-94.792 to 110.526] | -72.07 [-74.727 to -55.556] | -90.59 [-95.489 to -54.545] | -90.59 [-96.390 to 0.000]
  Cycle 3 Day 28: number analyzed (Participants) | 29 | 16 | 6 | 3 | 4 | 20
  Cycle 3 Day 28 | -80.00 [-95.833 to -53.191] | -96.06 [-98.193 to -37.085] | -66.27 [-87.847 to 184.211] | -79.63 [-83.718 to 21.484] | -66.60 [-96.992 to -45.455] | -90.45 [-97.611 to -53.191]
  Study Completion/Early Termination: number analyzed (Participants) | 41 | 15 | 17 | 5 | 4 | 19
  Study Completion/Early Termination | -49.31 [-85.444 to 2.941] | -87.00 [-95.725 to -14.925] | -45.44 [-52.500 to 37.500] | -75.09 [-93.911 to 1429.186] | -40.86 [-100.000 to 200.000] | -87.00 [-95.122 to 8.696]

19. Secondary Outcome: Absolute Change From Baseline in Measurements of T-cell Populations
Description: Actual change from baseline will be summarized descriptively by visit for the pharmacodynamic parameter: T-cell populations
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: 10^6 cells/L
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 71 | 26 | 30 | 9 | 6 | 32
10^6 cells/L
  Cycle 1 Day 8: number analyzed (Participants) | 64 | 24 | 27 | 8 | 5 | 29
  Cycle 1 Day 8 | 41.00 [-3.460 to 89.000] | 12.38 [-103.000 to 162.000] | 89.00 [46.000 to 260.000] | -55.92 [-219.000 to 600.000] | 16.00 [-1119.000 to 269.000] | 16.00 [-98.000 to 85.000]
  Cycle 1 Day 15: number analyzed (Participants) | 65 | 26 | 27 | 7 | 5 | 31
  Cycle 1 Day 15 | 12.00 [-67.000 to 80.000] | 3.00 [-301.000 to 123.000] | 28.00 [-43.000 to 196.000] | -22.00 [-193.000 to 1042.000] | -94.00 [-1011.000 to 526.000] | -19.00 [-297.790 to 110.000]
  Cycle 1 Day 22: number analyzed (Participants) | 61 | 23 | 26 | 7 | 5 | 28
  Cycle 1 Day 22 | -10.00 [-70.880 to 34.000] | -31.00 [-180.000 to 34.000] | 26.00 [-114.000 to 184.000] | -3.00 [-452.000 to 1129.500] | -41.00 [-252.000 to 71.000] | -36.00 [-180.000 to 26.000]
  Cycle 2 Day 1: number analyzed (Participants) | 58 | 24 | 24 | 5 | 5 | 29
  Cycle 2 Day 1 | 17.50 [-100.000 to 61.000] | -26.00 [-190.000 to 152.000] | 42.50 [-105.000 to 94.000] | -96.00 [-531.110 to 127.610] | -40.00 [-537.000 to 844.000] | -40.00 [-137.000 to 111.000]
  Cycle 2 Day 15: number analyzed (Participants) | 53 | 20 | 22 | 7 | 4 | 24
  Cycle 2 Day 15 | 88.00 [-9.000 to 152.000] | 59.98 [-117.000 to 153.000] | 72.00 [-115.000 to 184.000] | 164.00 [-9.000 to 719.030] | 54.50 [-28.000 to 422.000] | 59.98 [-72.000 to 153.000]
  Cycle 2 Day 28: number analyzed (Participants) | 48 | 21 | 18 | 5 | 4 | 25
  Cycle 2 Day 28 | 99.00 [-17.000 to 250.000] | 32.87 [-120.800 to 286.000] | 176.64 [-142.000 to 386.000] | 133.00 [39.320 to 1051.410] | 108.00 [-103.000 to 365.000] | 38.00 [-69.000 to 259.000]
  Cycle 3 Day 1: number analyzed (Participants) | 33 | 17 | 9 | 3 | 4 | 21
  Cycle 3 Day 1 | 58.00 [-69.000 to 158.500] | 45.00 [-140.000 to 267.000] | 115.00 [-100.000 to 222.700] | 174.00 [96.000 to 889.090] | -32.00 [-203.000 to 90.000] | -4.00 [-140.000 to 158.500]
  Cycle 3 Day 15: number analyzed (Participants) | 30 | 16 | 8 | 3 | 3 | 19
  Cycle 3 Day 15 | 110.00 [-27.000 to 318.000] | 94.00 [-111.930 to 383.000] | 203.50 [-517.000 to 462.000] | 599.00 [143.000 to 770.010] | -27.00 [-212.000 to 112.000] | 80.00 [-111.930 to 213.000]
  Cycle 3 Day 28: number analyzed (Participants) | 33 | 18 | 8 | 3 | 4 | 22
  Cycle 3 Day 28 | 102.45 [-40.000 to 243.000] | 72.23 [-110.000 to 448.000] | 198.31 [-403.000 to 696.000] | 131.00 [-131.000 to 1279.070] | 72.50 [-78.000 to 366.000] | 72.50 [-40.000 to 366.000]
  Study Completion/Early Termination: number analyzed (Participants) | 44 | 17 | 18 | 5 | 4 | 21
  Study Completion/Early Termination | -57.50 [-137.000 to 144.000] | -104.00 [-224.000 to 228.470] | -84.00 [-305.000 to 139.000] | 165.00 [-174.000 to 361.170] | 361.50 [-1079.000 to 2592.000] | -55.00 [-224.000 to 411.000]

20. Secondary Outcome: Percent Change From Baseline in Measurements of T-cell Populations
Description: Relative change from baseline will be summarized descriptively by visit for the pharmacodynamic parameter: T-cell populations
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 71 | 26 | 30 | 9 | 6 | 32
percentage change from baseline
  Cycle 1 Day 8: number analyzed (Participants) | 64 | 24 | 27 | 8 | 5 | 29
  Cycle 1 Day 8 | 7.28 [-0.394 to 16.991] | 1.59 [-8.906 to 18.456] | 17.07 [10.242 to 37.132] | -7.26 [-35.371 to 83.565] | 5.11 [-47.800 to 16.205] | 1.60 [-8.906 to 15.018]
  Cycle 1 Day 15: number analyzed (Participants) | 65 | 26 | 27 | 7 | 5 | 31
  Cycle 1 Day 15 | 1.75 [-9.999 to 12.312] | 1.25 [-17.200 to 14.604] | 8.81 [-15.314 to 44.118] | -4.01 [-26.187 to 145.125] | -17.49 [-43.187 to 31.687] | -1.99 [-17.491 to 12.312]
  Cycle 1 Day 22: number analyzed (Participants) | 61 | 23 | 26 | 7 | 5 | 28
  Cycle 1 Day 22 | -1.63 [-10.213 to 6.436] | -1.83 [-13.413 to 6.436] | 5.62 [-20.394 to 39.280] | -0.41 [-82.332 to 168.088] | -10.76 [-38.693 to 22.684] | -3.17 [-13.012 to 4.361]
  Cycle 2 Day 1: number analyzed (Participants) | 58 | 24 | 24 | 5 | 5 | 29
  Cycle 2 Day 1 | 2.93 [-12.484 to 12.025] | -1.63 [-17.286 to 14.765] | 10.38 [-7.023 to 20.524] | -12.48 [-76.529 to 14.538] | -12.78 [-38.701 to 50.843] | -2.36 [-17.286 to 14.765]
  Cycle 2 Day 15: number analyzed (Participants) | 53 | 20 | 22 | 7 | 4 | 24
  Cycle 2 Day 15 | 10.39 [-1.170 to 22.944] | 7.34 [-11.716 to 23.043] | 15.35 [-11.358 to 38.971] | 12.25 [-1.170 to 107.003] | 3.46 [-7.910 to 18.026] | 6.82 [-7.910 to 22.944]
  Cycle 2 Day 28: number analyzed (Participants) | 48 | 21 | 18 | 5 | 4 | 25
  Cycle 2 Day 28 | 9.91 [-3.321 to 30.339] | 5.96 [-8.938 to 29.916] | 36.51 [-10.132 to 73.662] | 20.58 [5.666 to 156.467] | 17.52 [-29.096 to 64.488] | 7.64 [-7.240 to 27.157]
  Cycle 3 Day 1: number analyzed (Participants) | 33 | 17 | 9 | 3 | 4 | 21
  Cycle 3 Day 1 | 12.99 [-6.114 to 23.810] | 9.60 [-9.799 to 27.929] | 18.67 [-7.159 to 43.226] | 17.49 [12.995 to 132.311] | -2.37 [-35.866 to 28.754] | -1.13 [-9.799 to 27.929]
  Cycle 3 Day 15: number analyzed (Participants) | 30 | 16 | 8 | 3 | 3 | 19
  Cycle 3 Day 15 | 20.09 [-7.627 to 34.934] | 9.57 [-12.210 to 34.934] | 20.66 [-14.130 to 100.873] | 44.73 [26.047 to 114.590] | -7.63 [-37.456 to 35.783] | 6.38 [-12.210 to 34.934]
  Cycle 3 Day 28: number analyzed (Participants) | 33 | 18 | 8 | 3 | 4 | 22
  Cycle 3 Day 28 | 17.34 [-9.783 to 26.905] | 11.37 [-13.423 to 33.794] | 21.90 [-18.260 to 151.965] | 23.86 [-9.783 to 190.346] | 17.10 [-13.781 to 32.588] | 14.15 [-11.156 to 32.588]
  Study Completion/Early Termination: number analyzed (Participants) | 44 | 17 | 18 | 5 | 4 | 21
  Study Completion/Early Termination | -8.07 [-14.994 to 26.912] | -12.80 [-18.456 to 29.129] | -8.07 [-42.093 to 32.548] | 12.32 [-31.694 to 52.042] | 28.31 [-65.000 to 457.951] | -12.21 [-18.456 to 29.712]

21. Secondary Outcome: Absolute Change From Baseline in Measurements of NK Cell Populations
Description: Actual change from baseline will be summarized descriptively by visit for the pharmacodynamic parameter: NK cell populations
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: 10^6 cells/L
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 71 | 26 | 30 | 9 | 6 | 32
10^6 cells/L
  Cycle 1 Day 8: number analyzed (Participants) | 64 | 24 | 27 | 8 | 5 | 29
  Cycle 1 Day 8 | -2.20 [-21.000 to 15.000] | -20.00 [-38.000 to 15.000] | 20.00 [-10.000 to 41.000] | -59.50 [-113.860 to 6.570] | 8.00 [-300.000 to 70.000] | -20.00 [-38.000 to 15.000]
  Cycle 1 Day 15: number analyzed (Participants) | 65 | 26 | 27 | 7 | 5 | 31
  Cycle 1 Day 15 | -23.00 [-43.000 to 11.000] | -36.99 [-67.000 to 28.090] | -4.00 [-26.250 to 23.000] | -33.00 [-216.000 to 117.000] | -79.00 [-211.000 to 66.000] | -38.97 [-73.000 to 20.000]
  Cycle 1 Day 22: number analyzed (Participants) | 61 | 23 | 26 | 7 | 5 | 28
  Cycle 1 Day 22 | -18.00 [-38.000 to 7.550] | -28.00 [-48.000 to 7.550] | 27.06 [-24.000 to 71.000] | -133.68 [-248.000 to -6.440] | -60.00 [-345.000 to 42.000] | -30.00 [-60.000 to 6.000]
  Cycle 2 Day 1: number analyzed (Participants) | 58 | 24 | 24 | 5 | 5 | 29
  Cycle 2 Day 1 | -16.32 [-33.000 to 9.890] | -11.01 [-39.730 to 21.000] | -21.31 [-37.000 to 19.000] | -64.00 [-249.000 to 556.030] | -1.00 [-146.000 to 135.000] | -7.00 [-31.000 to 21.000]
  Cycle 2 Day 15: number analyzed (Participants) | 53 | 20 | 22 | 7 | 4 | 24
  Cycle 2 Day 15 | -19.00 [-32.000 to 16.800] | 6.00 [-29.000 to 35.000] | -14.00 [-47.450 to 72.000] | -116.65 [-144.000 to 199.590] | -51.50 [-231.000 to 5.000] | -7.00 [-29.000 to 27.370]
  Cycle 2 Day 28: number analyzed (Participants) | 48 | 21 | 18 | 5 | 4 | 25
  Cycle 2 Day 28 | -1.00 [-18.000 to 51.000] | -3.00 [-23.980 to 48.000] | 52.00 [-31.000 to 76.000] | -93.00 [-181.270 to 10.430] | 9.50 [-260.000 to 245.000] | -3.00 [-23.980 to 48.000]
  Cycle 3 Day 1: number analyzed (Participants) | 33 | 17 | 9 | 3 | 4 | 21
  Cycle 3 Day 1 | -23.00 [-66.000 to -3.000] | -10.00 [-37.000 to 10.740] | -11.76 [-75.000 to 58.000] | -104.00 [-111.260 to -66.000] | -80.00 [-378.000 to 189.000] | -23.00 [-66.000 to 10.740]
  Cycle 3 Day 15: number analyzed (Participants) | 30 | 16 | 8 | 3 | 3 | 19
  Cycle 3 Day 15 | -33.00 [-70.000 to -2.000] | -27.50 [-63.000 to 41.000] | -46.00 [-75.800 to 158.000] | -99.00 [-153.310 to -24.000] | -84.00 [-97.000 to 88.000] | -29.00 [-67.000 to 41.000]
  Cycle 3 Day 28: number analyzed (Participants) | 33 | 18 | 8 | 3 | 4 | 22
  Cycle 3 Day 28 | -15.00 [-32.000 to 11.000] | -5.66 [-28.000 to 51.000] | 0.62 [-58.000 to 108.000] | -70.00 [-115.000 to -57.020] | -13.50 [-93.000 to 103.000] | -13.50 [-28.000 to 51.000]
  Study Completion/Early Termination: number analyzed (Participants) | 43 | 16 | 18 | 5 | 4 | 20
  Study Completion/Early Termination | -11.00 [-35.000 to 2.000] | -11.50 [-35.000 to -2.000] | -20.74 [-181.990 to 13.260] | 1.15 [-242.000 to 151.000] | 22.00 [-463.000 to 1924.000] | -9.00 [-35.000 to 8.000]

22. Secondary Outcome: Percent Change From Baseline in Measurements of NK Cell Populations
Description: Relative change from baseline will be summarized descriptively by visit for the pharmacodynamic parameter: NK cell populations
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 71 | 26 | 30 | 9 | 6 | 32
percentage change from baseline
  Cycle 1 Day 8: number analyzed (Participants) | 64 | 24 | 27 | 8 | 5 | 29
  Cycle 1 Day 8 | -1.62 [-18.261 to 11.429] | -11.58 [-23.789 to 6.122] | 13.16 [-16.393 to 36.190] | -32.20 [-43.326 to 3.990] | 13.79 [-48.940 to 194.444] | -8.66 [-23.789 to 13.793]
  Cycle 1 Day 15: number analyzed (Participants) | 65 | 26 | 27 | 7 | 5 | 31
  Cycle 1 Day 15 | -18.85 [-24.046 to 11.364] | -22.39 [-29.630 to 17.918] | -1.14 [-21.078 to 33.333] | -25.78 [-50.781 to 103.540] | -32.11 [-49.421 to 183.333] | -22.45 [-32.114 to 17.918]
  Cycle 1 Day 22: number analyzed (Participants) | 61 | 23 | 26 | 7 | 5 | 28
  Cycle 1 Day 22 | -13.38 [-29.688 to 3.027] | -13.38 [-39.053 to 3.027] | 18.16 [-36.667 to 69.880] | -50.87 [-78.000 to -4.347] | -36.21 [-56.281 to 116.667] | -14.59 [-39.053 to 2.597]
  Cycle 2 Day 1: number analyzed (Participants) | 58 | 24 | 24 | 5 | 5 | 29
  Cycle 2 Day 1 | -11.17 [-23.478 to 5.634] | -8.03 [-25.573 to 11.896] | -14.97 [-24.740 to 17.297] | -50.00 [-53.667 to 337.684] | -0.16 [-56.371 to 141.667] | -6.48 [-25.573 to 11.896]
  Cycle 2 Day 15: number analyzed (Participants) | 53 | 20 | 22 | 7 | 4 | 24
  Cycle 2 Day 15 | -8.11 [-22.467 to 20.314] | 9.03 [-22.467 to 22.727] | -7.13 [-31.429 to 60.000] | -41.00 [-56.250 to 134.731] | -20.08 [-37.684 to 8.621] | -1.51 [-22.467 to 20.370]
  Cycle 2 Day 28: number analyzed (Participants) | 48 | 21 | 18 | 5 | 4 | 25
  Cycle 2 Day 28 | -1.92 [-14.762 to 29.730] | -4.23 [-15.909 to 19.592] | 32.57 [-14.762 to 73.729] | -48.44 [-68.976 to 6.334] | 35.32 [-42.414 to 261.111] | -4.23 [-15.909 to 19.592]
  Cycle 3 Day 1: number analyzed (Participants) | 33 | 17 | 9 | 3 | 4 | 21
  Cycle 3 Day 1 | -14.08 [-26.866 to -1.115] | -12.83 [-25.191 to 12.987] | -8.33 [-35.545 to 50.000] | -42.34 [-51.563 to -34.667] | -31.97 [-61.664 to 525.000] | -13.22 [-26.866 to 12.987]
  Cycle 3 Day 15: number analyzed (Participants) | 30 | 16 | 8 | 3 | 3 | 19
  Cycle 3 Day 15 | -20.13 [-38.253 to -1.136] | -17.76 [-40.845 to 18.062] | -16.17 [-39.336 to 124.576] | -33.00 [-58.337 to -18.750] | -32.43 [-39.431 to 244.444] | -20.37 [-39.431 to 18.062]
  Cycle 3 Day 28: number analyzed (Participants) | 33 | 18 | 8 | 3 | 4 | 22
  Cycle 3 Day 28 | -6.10 [-21.697 to 17.000] | -2.72 [-24.426 to 19.872] | 1.78 [-28.409 to 91.525] | -38.33 [-54.688 to -21.697] | -5.37 [-15.171 to 286.111] | -5.37 [-18.182 to 19.872]
  Study Completion/Early Termination: number analyzed (Participants) | 43 | 16 | 18 | 5 | 4 | 20
  Study Completion/Early Termination | -11.01 [-28.906 to 6.667] | -11.06 [-28.333 to -0.866] | -23.94 [-62.726 to 16.667] | 0.78 [-80.667 to 86.979] | 42.15 [-75.530 to 782.114] | -10.49 [-28.333 to 22.222]

23. Secondary Outcome: Evaluation of AEs Stratified by Baseline CD19 Expression on Malignant Lymphoma Cells
Description: Incidence of AEs as stratified by presence of CD19 on malignant lymphoma cells detected by tumor biopsy/aspirate during Screening
Time Frame: From first dose until 30 days after last dose of MOR00208, up to 8.5 years
Population: Per pre-specified analysis plan, if CD19 expression on tumor cells was able to be measured in less than 15% of the ITT population at screening, the stratification analyses by baseline CD19 expression (as planned in the protocol) would not be performed. It was not possible to measure CD19 expression in sufficient cases for such an analysis to be meaningful.
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Evaluation of ORR Stratified by Baseline CD19 Expression on Malignant Lymphoma Cells
Description: The analysis of the primary endpoint (ORR) will additionally be stratified by presence of CD19 on malignant lymphoma cells detected by tumor biopsy/aspirate during Screening
Time Frame: From first dose until Follow-up Visit 12, up to 4.5 years
Population: as for outcome 23
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Evaluation of AEs Stratified by FcγRIIa Polymorphism
Description: Incidence of AEs as stratified by FcγRIIa polymorphism subgroups (genotypes HH, HR, or RR)
Time Frame: From first dose until 30 days after last dose of MOR00208, up to 8.5 years
Population: Genotyping for FcγRIIa and FcγRIIIa polymorphisms was performed for patients who consented to an optional mucosal cheek swab. Per pre-specified analysis plan, statistical summaries are provided overall, by NHL subtype, and for the combined group comprising FL patients + other iNHL patients.
Measure: Number; unit: adverse events
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 74 | 25 | 32 | 10 | 7 | 32
adverse events
  Genotype HH | 210 | 64 | 109 | 29 | 8 | 72
  Genotype HR | 188 | 83 | 51 | 6 | 48 | 131
  Genotype RR | 61 | 5 | 44 | 4 | 8 | 13

26. Secondary Outcome: Evaluation of AEs Stratified by FcγRIIIa Polymorphism
Description: Incidence of AEs as stratified by FcγRIIIa polymorphism subgroups (genotypes FF, FV, or VV)
Time Frame: From first dose until 30 days after last dose of MOR00208, up to 8.5 years
Population: as for outcome 25
Measure: Number; unit: adverse events
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 74 | 25 | 32 | 10 | 7 | 32
adverse events
  Genotype FF | 110 | 51 | 59 | 0 | 0 | 51
  Genotype FV | 149 | 75 | 33 | 33 | 8 | 83
  Genotype VV | 200 | 26 | 112 | 6 | 56 | 82

27. Secondary Outcome: Evaluation of ORR Stratified by FcγRIIa Polymorphism
Description: The analysis of the primary endpoint (ORR) will additionally be stratified by FcγRIIa polymorphism subgroups (genotypes HH, HR, or RR)
Time Frame: From first dose until Follow-up Visit 12, up to 4.5 years
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 74 | 25 | 32 | 10 | 7 | 32
Participants
  Genotype HH: number analyzed (Participants) | 24 | 9 | 11 | 3 | 1 | 10
  Genotype HH | 6 | 2 | 4 | 0 | 0 | 2
  Genotype HR: number analyzed (Participants) | 32 | 13 | 9 | 6 | 4 | 17
  Genotype HR | 8 | 3 | 3 | 0 | 2 | 5
  Genotype RR: number analyzed (Participants) | 18 | 3 | 12 | 1 | 2 | 5
  Genotype RR | 3 | 0 | 2 | 0 | 1 | 1

28. Secondary Outcome: Evaluation of ORR Stratified by FcγRIIIa Polymorphism
Description: The analysis of the primary endpoint (ORR) will additionally be stratified by FcγRIIIa polymorphism subgroups (genotypes FF, FV, or VV)
Time Frame: From first dose until Follow-up Visit 12, up to 4.5 years
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
Number analyzed (Participants) | 74 | 25 | 32 | 10 | 7 | 32
Participants
  Genotype FF: number analyzed (Participants) | 34 | 9 | 17 | 3 | 5 | 14
  Genotype FF | 10 | 1 | 6 | 0 | 3 | 4
  Genotype FV: number analyzed (Participants) | 30 | 12 | 10 | 6 | 2 | 14
  Genotype FV | 5 | 2 | 3 | 0 | 0 | 2
  Genotype VV: number analyzed (Participants) | 10 | 4 | 5 | 1 | 0 | 4
  Genotype VV | 2 | 2 | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from informed consent until 30 days after last dose of MOR00208, up to 8.5 years
Description: Patients were closely monitored for any kind of AE during the study. AEs were detected through physical examination, laboratory tests, or other assessments, or when volunteered by the patient in response to non-leading questioning during or between study visits. All SAEs are reported for the Safety Population, including events occurring prior to first dose of MOR00208. For non-serious AEs, only treatment-emergent events are reported (i.e., events occurring after first dose of MOR00208).
Arm/Group | Total | FL Subtype | DLBCL Subtype | MCL Subtype | Other iNHL | FL + Other iNHL
All-Cause Mortality (participants affected / at risk) | 9/92 | 1/34 | 6/35 | 2/12 | 0/11 | 1/45
Serious Adverse Events (participants affected / at risk) | 30/92 | 7/34 | 18/35 | 2/12 | 3/11 | 10/45
Other Adverse Events (participants affected / at risk) | 77/92 | 27/34 | 31/35 | 9/12 | 10/11 | 37/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=92) | FL Subtype (N=34) | DLBCL Subtype (N=35) | MCL Subtype (N=12) | Other iNHL (N=11) | FL + Other iNHL (N=45)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (5) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 11 (12) | 2 (3) | 6 (6) | 2 (2) | 1 (1) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=92) | FL Subtype (N=34) | DLBCL Subtype (N=35) | MCL Subtype (N=12) | Other iNHL (N=11) | FL + Other iNHL (N=45)
Neutropenia (Blood and lymphatic system disorders) | 9 (12) | 2 (2) | 5 (8) | 1 (1) | 1 (1) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (14) | 0 (0) | 4 (12) | 1 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (9) | 2 (4) | 3 (4) | 1 (1) | 0 (0) | 2 (4)
Nausea (Gastrointestinal disorders) | 9 (11) | 4 (6) | 2 (2) | 0 (0) | 3 (3) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 2 (2) | 5 (6) | 0 (0) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (7) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 3 (3)
Fatigue (General disorders) | 8 (12) | 3 (5) | 3 (5) | 0 (0) | 2 (2) | 5 (7)
Oedema peripheral (General disorders) | 8 (9) | 2 (2) | 5 (5) | 1 (2) | 0 (0) | 2 (2)
Asthenia (General disorders) | 7 (9) | 3 (5) | 3 (3) | 1 (1) | 0 (0) | 3 (5)
Pyrexia (General disorders) | 5 (8) | 2 (2) | 1 (2) | 1 (1) | 1 (3) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 11 (14) | 7 (9) | 4 (5) | 0 (0) | 0 (0) | 7 (9)
Bronchitis (Infections and infestations) | 6 (8) | 1 (1) | 4 (5) | 0 (0) | 1 (2) | 2 (3)
Infusion-related reaction (Injury, poisoning and procedural complications) | 12 (15) | 4 (4) | 4 (6) | 2 (2) | 2 (3) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 10 (15) | 3 (3) | 4 (7) | 1 (1) | 2 (4) | 5 (7)
Dizziness (Nervous system disorders) | 9 (11) | 4 (4) | 2 (3) | 0 (0) | 3 (4) | 7 (8)
Insomnia (Psychiatric disorders) | 7 (8) | 4 (5) | 1 (1) | 2 (2) | 0 (0) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 2 (3) | 4 (8) | 0 (0) | 2 (3) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 0 (0) | 4 (6) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT01685008/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT01685008/SAP_001.pdf